CLINICAL TRIAL: NCT00971139
Title: Implementing Online Patient-Provider Communication Into Clinical Practice: Implementation Research
Brief Title: Implementing Online Patient-Provider Communication Into Clinical Practice
Acronym: OPPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Cornelia Ruland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCN191008/V50
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Cancer; Injury of Liver; Diabetes
Keywords: Online patient-provider communication; Organizational change; Symptom management
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Access to an OPPC service (Experimental): Access to an Internet-based messaging system where patients can ask questions and receive advice and support from care providers at the hospital and social counsellors
  Interventions: Behavioral: Access to an OPPC service
- Control group (No Intervention): Patients receiving usual care

INTERVENTIONS:
Behavioral: Access to an OPPC service — Access to an Internet-based messaging system where patients can ask questions and receive advice and support from care providers at the hospital and social counsellors
  Arms: Access to an OPPC service

SUMMARY:
This interdisciplinary, international collaboration study, including the the Norwegian Health Economy Administration (HELFO) will evaluate the effectiveness and real-world implementation of an online patient-provider communication (OPPC) service into rout ine practice. In Phase I we will identify patients and care providers requirements and organizational contexts, and use participatory design methods to adapt the OPPC service to users needs and the context of clinical practice. In Phase II we will offer study participants access to the OPPC service to understand implementation issues. In addition, we will conduct a pilot randomized clinical trial (usual care; OPPC) with 40 patients in each group that will be followed over 6 months.

DETAILED DESCRIPTION:
A rapidly growing research literature documents the importance of Health IT to improve communication between health care providers and their patients. Patient Internet portals and online patient-provider communication (OPPC) allow patients to stay connected with their care providers between clinical encounters, get help and advice for their symptoms and problems from home, better understand and manage their illness, and become more engaged in their care. Through better patient-provider partnerships and communication independent of face-to-face visits, health problems and side-effects of treatment can be more easily detected, prevented, and treated more quickly.

Therefore, the overall goal of this international collaboration study is to implement and evaluate the effects and use of a primarily nurse-administered OPPC service, including access to advice from physicians, dietitians and social counselors, as part of regular patient care; and using methods consistent with effectiveness research to bridge the gap between research evidence and translation into routine practice.

The specific aims of this study are twofold:

In Phase I the investigators will refine and implement an Internet-based OPPC service where patients can ask questions and receive advice and support from care providers and social counselors. The investigators will use participatory design methods to adapt an OPPC service to patients' needs; care providers' requirements; and the workflow and organizational and technical infrastructure of clinical practice by answering the following research questions:

What are the predisposing, enabling and reinforcing factors related to successful adoption, implementation and maintenance of the OPPC service such as: potential barriers to successful implementation; workflow adjustments, support and resources needed to implement and maintain the OPPC in daily clinical practice?

In Phase II we will offer study participants access to the OPPC service to understand implementation issues. In addition, we will conduct a pilot randomized clinical trial (usual care; OPPC) with 40 patients in each group that will be followed over 6 months to evaluate:

1. participation rate and OPPC use;
2. characteristics of high/low volume users, patient-caregiver communication and use patterns;
3. perceived usefulness and ease of use and
4. impacts on organizational change and interdisciplinary collaboration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age.
* Able to read/speak Norwegian and have Internet with secure access (BankID) at home.

Exclusion Criteria:

* Excluded are patients who have brain metastasis and patients with cerebral affection caused by the disease (e.g., encephalopathy) as this may affect their abilities to reliably report their symptoms.
* Excluded are also patients who receive a liver transplant indicated by cancer coli, as they participate in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Impacts of the OPPC service on organizational processes/organizational change such as care processes | End of study at 6 (8) months after last included patient

SECONDARY OUTCOMES:
Participation rate and OPPC use, perceived usefulness and ease of use | End of study at 6 (8) months after last included patient
Characteristics of high/low volume users, patient-caregiver communication and use patterns | End of study at 6 (8) months after last included patient

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ruland, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital - Rikshospitalet, Oslo, Norway

REFERENCES:
- [Background] Ruland CM, Borosund E, Varsi C. User requirements for a practice-integrated nurse-administered online communication service for cancer patients. Stud Health Technol Inform. 2009;146:221-5. PMID 19592838
- [Result] Varsi C, Gammon D, Wibe T, Ruland CM. Patients' reported reasons for non-use of an internet-based patient-provider communication service: qualitative interview study. J Med Internet Res. 2013 Nov 11;15(11):e246. doi: 10.2196/jmir.2683. PMID 24220233
- [Result] Wibe T, Helleso R, Varsi C, Ruland C, Ekstedt M. How does an online patient-nurse communication service meet the information needs of men with recently diagnosed testicular cancer? ISRN Nurs. 2012;2012:260975. doi: 10.5402/2012/260975. Epub 2012 Dec 4. PMID 23251816
- [Result] Wibe T, Ekstedt M, Helleso R, Varsi C, Ruland C. "You are not at all bothersome" - nurses' online communication with testicular cancer patients. NI 2012 (2012). 2012 Jun 23;2012:453. eCollection 2012. PMID 24199140
- [Derived] Varsi C, Ekstedt M, Gammon D, Ruland CM. Using the Consolidated Framework for Implementation Research to Identify Barriers and Facilitators for the Implementation of an Internet-Based Patient-Provider Communication Service in Five Settings: A Qualitative Study. J Med Internet Res. 2015 Nov 18;17(11):e262. doi: 10.2196/jmir.5091. PMID 26582138